CLINICAL TRIAL: NCT06509451
Title: Retention Rate of Giomer S-PRG Filler Containing Pit and Fissure Sealant Applied With or Without Etching by Using Split Mouth Technique: Randomized Clinical Trial
Brief Title: Retention Rate of Giomer Pit and Fissure Sealant Applied With or Without Etching
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar abd elmageed ahmed, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Giomer sealant with etching
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Caries Prevention
MeSH Terms: interventions — Pit and Fissure Sealants

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Giomer pit and fissure sealant without etching (Active Comparator): In the control group, an adequate amount of primer is applied onto the enamel surface with a microbrush, left undisturbed for 5 s and then air-dried gently to avoid blowing it away. Beautisealant is applied directly from the syringe into pits and fissures and light-cured for 10 s, according to the manufacturer's instructions.
  Interventions: Drug: Giomer pit and fissure sealant without etching
- Giomer pit and fissure sealant with etching (Experimental): In the intervention group, the same steps are done except for an additional initial etching step with phosphoric acid etching for 30 s (for the uncut enamel) before primer and sealant application.
  Interventions: Drug: Giomer pit and fissure sealant with etching

INTERVENTIONS:
Drug: Giomer pit and fissure sealant without etching — S-PRG filler containig pit and fissure sealant without etching step
  Other Names: Beautisealant without etching
  Arms: Giomer pit and fissure sealant without etching
Drug: Giomer pit and fissure sealant with etching — S-PRG filler containig pit and fissure sealant with etching step
  Other Names: Beautisealant with etching
  Arms: Giomer pit and fissure sealant with etching

SUMMARY:
The aim of this study is to evaluate the retention rate of Giomer S-PRG filler containing pit and fissure sealant applied with or without etching by using split mouth technique.with null hypothesis that Giomer S-PRG filler containing pit and fissure sealant applied either with or without etching will have the same retention rate.

DETAILED DESCRIPTION:
Study Settings:

The study will be carried out at the Conservative Dentistry Department, Faculty of Dentistry, Cairo University in Egypt. Ethical approval is taken from the Research Ethics Committee of the faculty of Dentistry, Cairo University. Signed informed consent is signed by each participant.

Recruitment:

Participants are recruited from the patients' flow at the clinics of the Conservative Dentistry Department of Faculty of Dentistry, Cairo university.

Eligibility Criteria:

Inclusion Criteria:

1. ICDAS score 0 or 1
2. Satisfactory oral hygiene
3. Normal salivary characteristics (consistency, pH, flow rate, buffering capacity)
4. Satisfactory cooperative behavior
5. Age between 15- 30 years old
6. Males or females
7. Subjects who signed informed consent

Exclusion Criteria:

1. ICDAS score > 1
2. Poor oral hygiene
3. Evidence of tempromandibular joint disorders or malocclusion

Materials used in this trial are the Giomer S-PRG filler containing pit and fissure sealant (Beautisealant) and its self etching primer (Beauisealant primer).

Control group:

In the control group, an adequate amount of primer will be applied onto the enamel surface with a microbrush, left undisturbed for 5 s and then air-dried gently to avoid blowing it away. Beautisealant will be applied directly from the syringe into pits and fissures and light-cured for 10 s, according to the manufacturer's instructions.

Intervention Group:

In the intervention group, the same steps will be done except for an additional initial etching step with phosphoric acid etching for 30 s (for the uncut enamel) before primer and sealant application.

Outcome Assessment:

The results of sealant retention were assessed according to the following criteria (Simonsen):

A complete retention B partial loss (B1, without caries; B2, with caries) C complete loss (C1, without caries; C2, with caries)

ELIGIBILITY:
Inclusion Criteria:

1. ICDAS score 0 or 1
2. Satisfactory oral hygiene
3. Normal salivary characteristics (consistency, pH, flow rate, buffering capacity)
4. Satisfactory cooperative behavior
5. Age between 15- 30 years old
6. Males or females
7. Subjects who signed informed consent

Exclusion Criteria:

1. ICDAS score > 1
2. Poor oral hygiene
3. Evidence of tempromandibular joint disorders or malocclusion

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
retention rate | 3 months, 6months , 1 year
  To assess the sealant retention rate either total retention, partial loss or total loss

CONTACTS AND LOCATIONS:
Overall Officials: Cairo, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry, cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elmokanen MA, Gad HMA. Retention rate of giomer S-PRG filler containing pit and fissure sealant applied with or without etching: a randomized clinical trial. BMC Oral Health. 2024 Nov 7;24(1):1356. doi: 10.1186/s12903-024-05096-7. PMID 39511504